CLINICAL TRIAL: NCT04862637
Title: Using High Resolution Impedance Manometry (HRIM) Combined With Videofluoroscopic Swallow Study (VFSS) to Investigate the Changes of Swallowing Function in Oral Cancer Patients
Brief Title: Detecting the Changes of Swallowing Function in Oral Cancer Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202101035RIND
Record Dates: First submitted 2021-04-21; First posted 2021-04-28 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Swallowing Function
Keywords: dysphagia; swallowing
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The evidence of swallowing changes in oral cancer patients is still limited. This study aimed to investigated the swallowing changes in these patients by using the videofluoroscopy (VFSS) and high resolution impedance manometry (HRIM).

DETAILED DESCRIPTION:
Objective: to investigated the swallowing changes in oral cancer patients by using the videofluoroscopy (VFSS) and high resolution impedance manometry (HRIM).

Methods: 1. patients are fulfilled tongue cancer diagnosis; 2.they will undergo VFSS and HRIM examinations before or after surgery if they experience discomfort while swallowing.

ELIGIBILITY:
Inclusion Criteria:

* patients elective received oral cancer surgery

Exclusion Criteria:

* 1. patients had major underlying disease, ex: heart, brain, lung, liver disease
* 2. coagulopathy
* 3.pregnancy
* 4. the patients could not have good compliance

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with the diagnosis of oral cancer
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Bolus presence time | 15 minutes during the examination
  Lower value indicates shorter bolus presence in the pharynx

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
ethical concerns